CLINICAL TRIAL: NCT01107197
Title: Nutritional Support in Malnourished Pressure Ulcer Patients: the Oligoelement Sore Trial (OEST)
Brief Title: Nutritional Support in Pressure Ulcer Patients
Acronym: OEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Collaborators: Nutricia, Inc. (Industry)
Responsible Party: Principal Investigator, FEDERICO D'ANDREA, Director of Clinical Nutrition Unit, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 473/CE (Study n° CE 61/07)
Record Dates: First submitted 2010-04-15; First posted 2010-04-20 (Estimated); Results first posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-01

CONDITIONS: Pressure Ulcers
Keywords: Pressure ulcers; Healing; Malnutrition; Nutritional support; Micronutrients
MeSH Terms: conditions — Pressure Ulcer; Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isonitrogenous isocaloric formula (Active Comparator): Patients were given standard diet plus 2 bottles of an hypercaloric oral formula isonitrogenous isocaloric to the experimental one
  Interventions: Dietary Supplement: Control formula
- Enriched nutrition formula (Experimental): Patients were given standard diet plus 2 bottles of an hypercaloric oral formula enriched in arginine, zinc and antioxidant oligoelements
  Interventions: Dietary Supplement: Enriched nutrition formula

INTERVENTIONS:
Dietary Supplement: Enriched nutrition formula — oral formula enriched in arginine, zinc and antioxidant oligoelements
  Other Names: Cubitan (NUTRICIA Italia)
  Arms: Enriched nutrition formula
Dietary Supplement: Control formula — Isonitrogenous isocaloric oral formula
  Arms: Isonitrogenous isocaloric formula

SUMMARY:
Pressure ulcers are frequently associated with malnutrition. Previous studies have reported that nutritional support can improve the healing rate of pressure ulcers but no attention has been clearly given to the nutritional status of the patient treated. Moreover, other investigators have suggested the additional healing power of some nutrients. Unfortunately, previous results have been unpowered by small sample size, poor monitoring of compliance to treatments and the confounding effect of other nutrients. The investigators aimed to test the effect and additional benefits of several micronutrients delivered through oral nutritional support on the healing rate of pressure ulcers in malnourished patients.

ELIGIBILITY:
Inclusion Criteria:

* patient or legal guardian or caregiver consent
* stage II, III or IV pressure ulcers
* malnutrition (as defined by low body mass index and/or unintentional weight loss and/or low serum albumin and/or reduced food intake [<60% of total daily estimated requirements])
* patients who can drink supplements
* home-care or long-term care

Exclusion Criteria:

* decompensated diabetes (HbA1C >7%)
* renal failure
* hepatic failure (Child B and C)
* current neoplastic disease
* any organ-failure
* immunosuppressive therapy
* connective tissue disease
* use of steroids
* obesity
* respiratory insufficiency (COPD)
* anemia (haemoglobin <10g/dL)
* previous neoplastic disease (<1 year since last treatment CT or RT)
* infected wounds
* cellulitis, sepsis or osteomyelitis
* poor tolerance to sip feeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Federico D'Andrea, MD, Principal Investigator — Azienda Ospedaliero Universitaria Maggiore della Carita
Locations (1):
- Azienda Ospedaliero Universitaria Maggiore della Carita, Novara, Italy

REFERENCES:
- [Background] Cereda E, Gini A, Pedrolli C, Vanotti A. Disease-specific, versus standard, nutritional support for the treatment of pressure ulcers in institutionalized older adults: a randomized controlled trial. J Am Geriatr Soc. 2009 Aug;57(8):1395-402. doi: 10.1111/j.1532-5415.2009.02351.x. Epub 2009 Jun 25. PMID 19563522
- [Background] Benati G, Delvecchio S, Cilla D, Pedone V. Impact on pressure ulcer healing of an arginine-enriched nutritional solution in patients with severe cognitive impairment. Arch Gerontol Geriatr Suppl. 2001;7:43-7. doi: 10.1016/s0167-4943(01)00120-0. No abstract available. PMID 11431045
- [Background] Frias Soriano L, Lage Vazquez MA, Maristany CP, Xandri Graupera JM, Wouters-Wesseling W, Wagenaar L. The effectiveness of oral nutritional supplementation in the healing of pressure ulcers. J Wound Care. 2004 Sep;13(8):319-22. doi: 10.12968/jowc.2004.13.8.26654. PMID 15469215
- [Background] Heyman H, Van De Looverbosch DE, Meijer EP, Schols JM. Benefits of an oral nutritional supplement on pressure ulcer healing in long-term care residents. J Wound Care. 2008 Nov;17(11):476-8, 480. doi: 10.12968/jowc.2008.17.11.31475. PMID 18978686
- [Background] van Anholt RD, Sobotka L, Meijer EP, Heyman H, Groen HW, Topinkova E, van Leen M, Schols JM. Specific nutritional support accelerates pressure ulcer healing and reduces wound care intensity in non-malnourished patients. Nutrition. 2010 Sep;26(9):867-72. doi: 10.1016/j.nut.2010.05.009. Epub 2010 Jul 3. PMID 20598855
- [Derived] Cereda E, Klersy C, Serioli M, Crespi A, D'Andrea F; OligoElement Sore Trial Study Group. A nutritional formula enriched with arginine, zinc, and antioxidants for the healing of pressure ulcers: a randomized trial. Ann Intern Med. 2015 Feb 3;162(3):167-74. doi: 10.7326/M14-0696. PMID 25643304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants: patients (long-term care residents or subjects at home care services) with stage 2, 3 or 4 pressure ulcer.
  Estimated recruitment (sample size): 220 patients. Patients recruited and randomized to interventionas: 200 patients. The recruitment was stopped when at least 64 patients per treatment arm were available for analyses.
Groups:
- Isonitrogenous Isocaloric Formula: Patients were given standard diet plus 2 bottles/day (200 mL each; in 4 boluses [100 mL each] spread throughout the day) of an hypercaloric oral formula isonitrogenous isocaloric to the experimental one for 8 weeks
  Control formula : Isonitrogenous isocaloric oral formula
- Enriched Nutrition Formula: Patients were given standard diet plus two bottles/day (400 mL) of an hypercaloric oral formula enriched in arginine, zinc and antioxidant oligoelements for 8 weeks
  Enriched nutrition formula : oral formula enriched in arginine, zinc and antioxidant oligoelements
Period: Overall Study
Arm/Group | Isonitrogenous Isocaloric Formula | Enriched Nutrition Formula
Started | 99 | 101
Completed | 79 (Included in intention-to-treat efficacy analyses (per-protocol analyses were based on 67 patients )) | 78 (Included in intention-to-treat efficacy analyses (per-protocol analyses were based on 64 patients ))
Not Completed | 20 | 23
Not completed — Death | 12 | 10
Not completed — Lost to Follow-up | 5 | 8
Not completed — Withdrawal by Subject | 3 | 5

BASELINE CHARACTERISTICS:
Population: Principal analysis were conducted according to the intention-to-treat (ITT) principle. ITT analyses were based on 157 patients. All patients who have been assessed at baseline and at least at 4 weeks will be included in the ITT population.
Groups:
- Enriched Nutrition Formula: Patients were given standard diet plus two brick of an hypercaloric oral formula enriched in arginine, zinc and antioxidant oligoelements
  Enriched nutrition formula : oral formula enriched in arginine, zinc and antioxidant oligoelements
- Isonitrogenous Isocaloric Formula: Patients were given standard diet plus 2 bricks of an hypercaloric oral formula isonitrogenous isocaloric to the experimental one
  Control formula : Isonitrogenous isocaloric oral formula
- Total: Total of all reporting groups
Arm/Group | Enriched Nutrition Formula | Isonitrogenous Isocaloric Formula | Total
Number analyzed (Participants) | 78 | 79 | 157
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 73 | 75 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.6 (11.4) | 81.2 (11.3) | 80.9 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 52 | 109
  Male | 21 | 27 | 48
Region of Enrollment [Number; unit: participants]
  Italy | 78 | 79 | 157

OUTCOME MEASURES:

1. Primary Outcome: Rate of Healing
Description: healing is defined as reduction in ulcer area (the percentage of change)
Time Frame: 8 weeks of nutritional support (baseline and week 8)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Enriched Nutrition Formula | Isonitrogenous Isocaloric Formula
Number analyzed (Participants) | 78 | 79
percent change | 62.9 (29.1) | 43.4 (33.5)

2. Secondary Outcome: Rate of Healing
Description: reduction in ulcer area >=40%
Time Frame: 8 weeks of nutritional support (baseline and week 8)
Measure: Number; unit: participants
Arm/Group | Enriched Nutrition Formula | Isonitrogenous Isocaloric Formula
Number analyzed (Participants) | 78 | 79
participants | 57 | 41

3. Secondary Outcome: Rate of Healing
Description: complete healing
Time Frame: 8 weeks of nutritional support (baseline and week 8)
Measure: Number; unit: participants
Arm/Group | Enriched Nutrition Formula | Isonitrogenous Isocaloric Formula
Number analyzed (Participants) | 78 | 79
participants | 12 | 6

4. Secondary Outcome: Incidence of Infections
Description: defined as local (ulcer)
Time Frame: 8 weeks of nutritional support (baseline and week 8)
Measure: Number; unit: participants
Arm/Group | Enriched Nutrition Formula | Isonitrogenous Isocaloric Formula
Number analyzed (Participants) | 78 | 79
participants | 9 | 14

5. Secondary Outcome: Cost-effectiveness
Description: Incremental cost-effectiveness ratio (ICER) was calculated by dividing the difference between total costs (active - control) by the difference in the mean reduction (%) of ulcer area. Costs are derived from oral nutritional supplements, dressings, antibiotics, PU swab sampling, nurse visits for wound dressing (according to their duration and cost per hour), medical consultations (unitary cost of the visit for prescription of antibiotic therapy).
Time Frame: 8 weeks of nutritional support (baseline and week 8)
Measure: Mean (Standard Deviation); unit: Euros
Arm/Group | Enriched Nutrition Formula | Isonitrogenous Isocaloric Formula
Number analyzed (Participants) | 78 | 79
Euros | 639 (213) | 689 (247)

6. Secondary Outcome: Dressings
Description: The number of dressings used throughout the intervention period
Time Frame: 8 weeks of nutritional support (baseline and week 8)
Measure: Mean (Standard Deviation); unit: dressings
Arm/Group | Enriched Nutrition Formula | Isonitrogenous Isocaloric Formula
Number analyzed (Participants) | 78 | 79
dressings | 31 (13) | 35 (13)

7. Secondary Outcome: the Percentage of Change in Area
Description: the reduction in ulcer area (%) observed at 4 weeks
Time Frame: 4 weeks of nutritional support (baseline and week 4)
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Enriched Nutrition Formula | Isonitrogenous Isocaloric Formula
Number analyzed (Participants) | 78 | 79
percent change | 29.3 [13.9 to 58.9] | 21.9 [5.6 to 38.1]

ADVERSE EVENTS:
Time Frame: 8 weeks of nutritional support
Description: Direct observation of the patient
Arm/Group | Enriched Nutrition Formula | Isonitrogenous Isocaloric Formula
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/99
Other Adverse Events (participants affected / at risk) | 0/101 | 0/99

LIMITATIONS AND CAVEATS:
Limited to specific settings: long-term care and home-care services Limited to malnourished patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No